CLINICAL TRIAL: NCT02225392
Title: Unravelling Targets of Therapy in Bronchial Thermoplasty in Severe Asthma
Acronym: TASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); The Netherlands Asthma Foundation (Other); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Prof. dr. J.T. Annema, Prof. dr. J.T. Annema, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL45394.018.13; 5.2.13.064 (Other Grant/Funding Number: Longfonds); 90713477 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2014-07-30; First posted 2014-08-26 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Asthma; Bronchial Asthma
Keywords: Bronchial thermoplasty; Severe asthma
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Delayed bronchial thermoplasty (Active Comparator): After randomisation they will wait for 25 weeks (control group) and then start with bronchial thermoplasty.
  Bronchial thermoplasty (BT) will be performed using the Alair system (Boston Scientific, USA). Patients will undergo 3 bronchoscopy procedures with BT at least 3 weeks apart. Treatment sessions are designed to address different lobes of the lung with the right lower lobe treated during the first bronchoscopy, the left lower lobe treated during the second bronchoscopy, and both the right and left upper lobes treated in the third and final bronchoscopy. The right middle lobe and proximal airways including RC2 are left untreated.
  Interventions: Procedure: Bronchial thermoplasty; Device: Alair system (Boston Scientific, USA)
- Immediate bronchial thermoplasty (Experimental): After randomisation they start immediate with bronchial thermoplasty treatment.
  Bronchial thermoplasty (BT) will be performed using the Alair system (Boston Scientific, USA). Patients will undergo 3 bronchoscopy procedures with BT at least 3 weeks apart. Treatment sessions are designed to address different lobes of the lung with the right lower lobe treated during the first bronchoscopy, the left lower lobe treated during the second bronchoscopy, and both the right and left upper lobes treated in the third and final bronchoscopy. The right middle lobe and proximal airways including RC2 are left untreated.
  Interventions: Procedure: Bronchial thermoplasty; Device: Alair system (Boston Scientific, USA)

INTERVENTIONS:
Procedure: Bronchial thermoplasty — Bronchial thermoplasty (BT) will be performed using the Alair system (Boston Scientific, USA). Patients will undergo 3 bronchoscopy procedures with BT at least 3 weeks apart. Treatment sessions are designed to address different lobes of the lung with the right lower lobe treated during the first bronchoscopy, the left lower lobe treated during the second bronchoscopy, and both the right and left upper lobes treated in the third and final bronchoscopy. The right middle lobe and proximal airways including RC2 are left untreated.
Device: Alair system (Boston Scientific, USA) — The alair system consist of a controller and a bastket catheter.

SUMMARY:
Approximately 5% of asthma patients suffer from severe asthma that is characterized by frequent asthma exacerbations resulting in significant morbidity and excessive utilisation of health care resources. Therefore, there is a strong need for improved therapeutic strategies for these patients. Insight in the pathogenesis and molecular pathways active in severe asthma is crucial to reach this goal.

Bronchial Thermoplasty (BT) is a novel, innovative device-based treatment of severe asthma that is based on local, radiofrequent energy delivery in larger airways during bronchoscopy.

Hypothesis:

BT-induced clinical improvement in severe asthma is a consequence of reduction in airway smooth muscle (ASM) mass and (contractile/immunomodulatory) function, inflammation, neural innervation and/or vascular integrity resulting in altered airway remodelling. BT target identification and severe asthma phenotyping are critical for improved patient selection for BT and fundamental to discover novel, specific signalling pathways active in severe asthma.

DETAILED DESCRIPTION:
This study has a two-fold purpose:

1. to unravel the targets of BT in severe asthma (how does it work?) which is fundamental for better patient selection (who benefits most?) and further improvement of BT technology and novel asthma therapy development (how to treat better?). These objectives can only be achieved by linking patient-reported outcomes to airway structure/function, which is the principal aim of the study proposed.
2. to investigate clinical outcome analyses

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 or greater and 65 or less
2. The diagnosis of asthma confirmed by at least one of the following as assessed at least once during the past 5 years before the study:

   * Reversibility to β2-agonists ≥12% predicted and ≥200ml after 400μg inhaled salbutamol or equivalent
   * Bronchial hyper-responsiveness to methacholine or histamine
   * Peak-flow variability of >20% over a period of 14 days
   * Fall in FEV1 >12% and >200ml when tapering treatment (ICS, oral steroid, LABA and/or LTRA).
3. Subject is taking regular maintenance medication (GINA step 4-5) for past 6 months that includes:

   * Inhaled corticosteroid at a dosage ≥500μg fluticasone equivalent per day AND
   * Long acting ß2-agonist at a dosage of ≥100μg per day salmeterol dose aerosol or equivalent).
4. Per protocol bronchial hyper-responsiveness to methacholine (PC20<4 mg/ml)
5. Other asthma medications are acceptable (such as Leukotriene modifiers, Theophylline, Omalizumab treatment (or discontinuation for at least 6 months) Systemic corticosteroid use (≤20mg/day prednisone equivalent))
6. Pre-bronchodilator FEV1 ≥50% predicted (stabilized on ICS/LABA) and post-bronchodilator FEV1 ≥60%
7. ACQ >1,5 for 2 weeks
8. Non-smoker for 1 year or more (former smoker ≤15 pack years)
9. Ability to undergo bronchoscopy and BT in the opinion of the investigator.
10. Ability and willingness to provide informed consent.
11. For women of childbearing potential: non pregnant, non-lactating, and agree to practice an adequate birth control method for the duration of the study.

Exclusion Criteria:

1. Asthma exacerbation during the prior 4 weeks.
2. Subject has 5 or more hospitalizations for exacerbations of asthma in the previous year or 1 or more ICU admission for mechanical or endotracheal intubation for asthma in the previous year.
3. Respiratory tract infection within past 4 weeks
4. Subject has a known sensitivity to medications required to perform bronchoscopy
5. Subject is using immunosuppressant therapy other than oral steroid therapy
6. Subject is on anticoagulant medication including anti-platelet agents.
7. Subject has bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 125,000/mm2 or known coagulopathy (INR >1.5).
8. Subject has other respiratory diseases including interstitial lung disease, emphysema, cystic fibrosis, mechanical upper airway obstruction, Churg-Strauss syndrome, and allergic bronchopulmonary aspergillosis (total IgE of >1000 Units/mL with positive specific IgE to aspergillus and evidence of central bronchiectasis).
9. Subject has segmental atelectasis, lobar consolidation, significant or unstable pulmonary infiltrate, or pneumothorax, confirmed on x-ray. Bronchiectasis on HR-CT-of the chest, both centrally or peripherally will be excluded.
10. Subject has clinically significant cardiovascular disease, including myocardial infarction, angina, cardiac dysrhythmia, conduction defect, cardiomyopathy, aortic aneurysm, or stroke at the discretion of the investigator
11. Subject has uncontrolled hypertension (>200mmHg systolic or >100mmHg diastolic pressure).
12. Subject uses an internal or external pacemaker or cardiac defibrillator.
13. Other chronic diseases that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation, e.g. liver, kidney, or nervous system
14. Current smokers, and a history of cigarette smoking with >15 pack years total
15. Use of investigative drugs or intervention trials in the 4 months prior to enrolment or during the duration of the study
16. Any condition or compliance issue which in the opinion of the investigator might interfere with participation inthe study
17. BMI >35
18. Pre-bronchodilator FEV1 <1.2L
19. Extreme coughing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
The change in airway smooth muscle (ASM) mass between immediate BT treated and the control group (N=20, randomized) | Baseline, week 25
  The change in ASM mass as determined by the percentage of ASM surface area in airway biopsies between:
  * the immediate BT group and
  * the delayed BT group = control group

SECONDARY OUTCOMES:
The change in ASM mass in airway biopsies before and after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 25 weeks
  Change in ASM mass in endobronchial biopsies before and after bronchial thermoplasty treatment
The change in structural airway remodelling after and during bronchial thermoplasty treatment | Baseline, week 25
  Optical Coherence Tomography (OCT)- and/or Radial Endobronchial ultrasound (rEBUS)-determined changes in structural airway remodelling.
The change in pre-and post bronchodilator FEV1 and related % reversibility between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in PC20 methacholine between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in Fraction of exhaled nitric oxide (FeNO) between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in asthma control questionnaire (ACQ) between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in - asthma related quality of life questionnaire (AQLQ) between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in health care utilization between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in rescue medication use between immediate BT treated and control group (N=20, randomized) | Baseline, 24 week
The change in inflammatory cell density/counts in biopsy, BAL and induced sputum between immediate BT treated and control group (N=20, randomized) | Baseline, 25 week
The change in pre-and post bronchodilator FEV1 and related % reversibility after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in PC20 methacholine after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in Fraction of exhaled nitric oxide (FeNO) after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in asthma control questionnaire (ACQ) after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in asthma related quality of life questionnaire (AQLQ) after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in health care utilization after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in rescue medication use after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 24 week
The change in inflammatory cell density/counts in biopsy, BAL and induced sputum before and after bronchial thermoplasty treatment (N=40, observational, before and after BT) | Baseline, 25 week

OTHER OUTCOMES:
The change in Airway-resistance (sRaw)/-conductance(sGaw)/-mechanics (forced oscillation technique (FOT)) parameters after bronchial thermoplasty treatment | Baseline, 24 weeks
The change in exhaled volatile organic compounds (VOCs) after bronchial thermoplasty treatment | Baseline, 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jouke T Annema, Prof. Dr., Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); P I Bonta, Dr, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (3):
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - University Medical Center Groningen, Groningen
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Wijsman PC, Goorsenberg AWM, Keijzer N, d'Hooghe JNS, Ten Hacken NHT, Shah PL, Weersink EJM, de Brito JM, de Souza Xavier Costa N, Mauad T, Nawijn MC, Vonk JM, Annema JT, Burgess JK, Bonta PI. Airway wall extracellular matrix changes induced by bronchial thermoplasty in severe asthma. J Allergy Clin Immunol. 2024 Feb;153(2):435-446.e4. doi: 10.1016/j.jaci.2023.09.035. Epub 2023 Oct 5. PMID 37805024
- [Derived] Goorsenberg AWM, d'Hooghe JNS, Slats AM, van den Aardweg JG, Annema JT, Bonta PI. Resistance of the respiratory system measured with forced oscillation technique (FOT) correlates with bronchial thermoplasty response. Respir Res. 2020 Feb 12;21(1):52. doi: 10.1186/s12931-020-1313-6. PMID 32050956
- [Derived] d'Hooghe JNS, Ten Hacken NHT, Weersink EJM, Sterk PJ, Annema JT, Bonta PI. Emerging understanding of the mechanism of action of Bronchial Thermoplasty in asthma. Pharmacol Ther. 2018 Jan;181:101-107. doi: 10.1016/j.pharmthera.2017.07.015. Epub 2017 Jul 27. PMID 28757156